CLINICAL TRIAL: NCT03219632
Title: Angiotensin Blocking Effect of Fimasartan on Hypertensive Cardiac Disease With Left Ventricular Hypertrophy Estimated by ECG: a Prospective, Multicenter, Observational Registry
Brief Title: Fimasartan on Hypertensive Cardiac Disease With Left Ventricular Hypertrophy Estimated by ECG
Status: Completed | Type: Observational
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Dong-Ju Choi, Professor, MD, PhD, Seoul National University Bundang Hospital
Other Study IDs: ACADEMY
Record Dates: First submitted 2017-07-12; First posted 2017-07-17 (Actual); Last update posted 2017-07-17 (Actual); Status verified 2017-07

CONDITIONS: Left Ventricular Hypertrophy; Hypertension
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Hypertension | interventions — fimasartan

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 1 Year
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Drug: Fimasartan — Fimasartan is a non-peptide angiotensin II receptor antagonist (ARB) used for the treatment of hypertension and heart failure.

SUMMARY:
Assess the efficacy of fimasartan on left ventricular hypertrophy in hypertensive patients

DETAILED DESCRIPTION:
Patients who were diagnosed with left ventricular hypertrophy (LVH) by ECG at the start of the study are followed up at 3-month intervals for 1 year.

Increase Fimasartan if blood pressure is not controlled.

ELIGIBILITY:
Inclusion Criteria:

* Patients who have been treated or not treated with hypertension from 20 to 80 years of age
* Patients with electrocardiographic left ventricular hypertrophy (In this study, we define left ventricular hypertrophy if one of the following two criteria is met)

  1. RaVL+SV3 > 20mm(M). 16mm(F)
  2. SV1+RV5 or RV6 > 35mm.
* Patients who are taking or expecting Fimasartan

Exclusion Criteria:

* Patients with unstable angina or myocardial infarction within 3 months
* Patients with clinically significant severe valve disease, congenital heart disease, peripheral vascular disease, cerebrovascular disease
* Clinically significant severe congestive heart failure patients
* Patients with renal dialysis
* Clinically significant renal disease patients
* Patients with clinically significant hepatic impairment
* Patients with a history of alcohol or substance abuse
* Patients with hypersensitivity to angiotensin-receptor blocker
* Patients needing angiotensin-receptor blocker drugs other than fimasartan
* For women, pregnancy, Patients who are breastfeeding or planning to become pregnant
* A person who is determined to be inappropriate by the Investigator
* Patients participating in other clinical trials

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Registered 319 people considering 30% dropout rate
Sampling Method: Non-Probability Sample
Enrollment: 72 (Actual)
Dates: Start 2012-06-05 (Actual); Primary Completion 2017-04-30 (Actual); Study Completion 2017-05-30 (Actual)

PRIMARY OUTCOMES:
The change in systolic and diastolic blood pressure, left ventricular hypertrophy in ECG (composite). | 1 year
  Measurements of changes in baseline at 12 months (change in systolic and diastolic blood pressure, left ventricular hypertrophy in ECG)

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Ju choi, Principal Investigator — Seoul National University Bundang Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Vakili BA, Okin PM, Devereux RB. Prognostic implications of left ventricular hypertrophy. Am Heart J. 2001 Mar;141(3):334-41. doi: 10.1067/mhj.2001.113218. PMID 11231428
- [Background] Katholi RE, Couri DM. Left ventricular hypertrophy: major risk factor in patients with hypertension: update and practical clinical applications. Int J Hypertens. 2011;2011:495349. doi: 10.4061/2011/495349. Epub 2011 Jun 30. PMID 21755036
- [Background] Sadoshima J, Izumo S. Molecular characterization of angiotensin II--induced hypertrophy of cardiac myocytes and hyperplasia of cardiac fibroblasts. Critical role of the AT1 receptor subtype. Circ Res. 1993 Sep;73(3):413-23. doi: 10.1161/01.res.73.3.413. PMID 8348686
- [Background] Okin PM, Devereux RB, Jern S, Kjeldsen SE, Julius S, Nieminen MS, Snapinn S, Harris KE, Aurup P, Edelman JM, Dahlof B; Losartan Intervention for Endpoint reduction in hypertension Study Investigations. Regression of electrocardiographic left ventricular hypertrophy by losartan versus atenolol: The Losartan Intervention for Endpoint reduction in Hypertension (LIFE) Study. Circulation. 2003 Aug 12;108(6):684-90. doi: 10.1161/01.CIR.0000083724.28630.C3. Epub 2003 Jul 28. PMID 12885747